A Multicenter, Open-Label, Randomized, Controlled Phase III Clinical
Study Comparing UTD2 Combined with Capecitabine to Capecitabine
Monotherapy as Adjuvant Therapy for Triple-Negative Early Breast
Cancer Patients Who Did Not Achieve Pathological Complete Response
After Neoadjuvant Therapy

| Sponsor | Fudan University Shanghai Cancer Center |
|---|---|
| Investigational | Utidelone Capsules (UTD2) |
| Product | |
| Study ID | BG02-T2401 |
| Study Title | A Multicenter, Open-Label, Randomized, Controlled Phase III Clinical |
| | Study Comparing UTD2 Combined with Capecitabine to Capecitabine |
| | Monotherapy as Adjuvant Therapy for Triple-Negative Early Breast Cancer |
| | Patients Who Did Not Achieve Pathological Complete Response After |
| | Neoadjuvant Therapy |
| Phase | Phase III |
| Phase III | Prof. Zhi-Min Shao |
| Number of | Approximately 39 centers |
| Sites | |
| Study | Triple-negative early breast cancer patients who did not achieve pCR after |
| Population | neoadjuvant therapy |
| Study<br>Objectives | <b>Primary Objective</b> To evaluate the 3-year invasive disease-free survival |
| | (IDFS) rate of UTD2 combined with capecitabine versus capecitabine |
| | monotherapy in adjuvant therapy for triple-negative early breast cancer |
| | patients who did not achieve pCR after neoadjuvant therapy. |
| | Secondary Objectives - Compare IDFS rates (3-year and 5-year), overall |
| | survival (OS) rates (3-year and 5-year), and safety profiles between the two |
| | arms. |
| | Exploratory Objectives - Identify predictive/prognostic biomarkers using |
| | tumor/adjacent tissues, blood, and stool samples. |
| | - Investigate molecular features associated with treatment response and |
| | tumor biology. |
| Endpoints | Primary Endpoint 3-year IDFS rate |
| | Secondary Endpoints 5-year IDFS rate, 3-year OS rate, 5-year OS rate, |
| | safety analysis (CTCAE v5.0) |
| | Translational Endpoints Biomarker discovery and correlation with |
| | disease status/treatment response. |

Design: Multicenter, open-label, randomized, controlled, superiority Phase III trial.

Sample Size: 440 patients (1:1 randomization: 220 in UTD2 + capecitabine arm; 220 in capecitabine monotherapy arm).

Stratification Factor: Postoperative pathological lymph node status (negative vs. positive).

Treatment Regimens:

## Study Design

Experimental Arm:

UTD2: 50 mg/m²/day orally on Days 1–5, repeated every 21 days for 2 years.

Capecitabine: 1000 mg/m² orally twice daily on Days 1–14, repeated every 21 days for 8 cycles.

Control Arm:

Capecitabine: Same dose and schedule as above.

Follow-up: Imaging every 6 months to assess disease recurrence.

# Inclusion Criteria

#### 1.Informed Consent and Compliance

The patient has fully understood this study and voluntarily signed the informed consent form, demonstrating the ability and willingness to comply with the study protocol-defined visits, treatment plans, laboratory tests, and other study procedures.

2.Age and Gender

Female patients aged 18 to 70 years old (inclusive) on the day of signing the informed consent.

3. Prior Neoadjuvant Chemotherapy without pCR

Received prior neoadjuvant chemotherapy containing anthracycline or taxane agents without achieving pathological complete response (pCR).

Neoadjuvant chemotherapy requirement: At least 4 completed cycles.

Non-pCR definition: Residual invasive carcinoma confirmed by pathology after primary tumor resection.

4. Surgical Resection

Underwent complete surgical resection (R0) with pathologically confirmed negative margins.

5. Triple-Negative Breast Cancer Confirmation

Post-resection tumor tissue confirmed as ER-negative, PR-negative, and

HER2-negative breast cancer by immunohistochemistry (IHC):

ER-negative: <1% expression by IHC.

PR-negative: <1% expression by IHC.

HER2-negative: IHC score of 0 or 1+, or 2+ with negative in situ hybridization (ISH) results.

6.Postoperative Treatment

No prior systemic anticancer therapy (excluding radiotherapy) after breast cancer surgery.

7.Performance Status

ECOG performance status of 0 to 1.

8. Hematological Criteria (within 1 week prior to enrollment)

Blood tests meet the following criteria (CTCAE v5.0  $\leq$  Grade 1, based on institutional laboratory standards):

White blood cell (WBC) count  $\geq 3.0 \times 10^{9}$ L.

Absolute neutrophil count (ANC)  $\geq 1.5 \times 10^{9}$ L.

Platelet (PLT) count  $\geq 100 \times 10^{9}$ /L.

Hemoglobin  $\geq 9.0 \text{ g/dL}$ .

No administration of recombinant human granulocyte colony-stimulating factor (rhG-CSF), blood products, or erythropoietin (EPO) within 14 days prior to enrollment.

9. Biochemical Criteria (within 1 week prior to enrollment)

Normal blood biochemistry (CTCAE v5.0  $\leq$  Grade 1, based on institutional laboratory standards):

Total bilirubin (TBIL)  $\leq 1.5 \times$  upper limit of normal (ULN).

Alanine aminotransferase (ALT)  $\leq 1.5 \times ULN$ .

Aspartate aminotransferase (AST)  $\leq 1.5 \times ULN$ .

Alkaline phosphatase (ALP)  $\leq 2.5 \times \text{ULN}$ .

Creatinine clearance (Ccr)  $\geq$  50 mL/min.

Contraception Requirements

Fertile patients must agree to use highly effective contraception (hormonal, barrier methods, or abstinence) with their partners during the trial and for at least 6 months after the last dose. Premenopausal female patients must have a

| | negative blood or urine pregnancy test before enrollment. |
|---|---|
| | 1.Stage IV metastatic breast cancer. |
| Exclusion<br>Criteria | 2.Bilateral breast cancer. |
| Cittoria | 3. History of other malignancies within the past 5 years, except for cured |
| | basal cell carcinoma of the skin, cervical carcinoma in situ, or papillary |
| | thyroid carcinoma. |
| | 4.Radiotherapy within 2 weeks prior to the first dose of the study drug. |
| | 5.Surgery within 2 weeks prior to the first dose of the study drug. |
| | 6.Prior treatment with utidelone or capecitabine, known hypersensitivity to |
| | utidelone, capecitabine, or fluoropyrimidines, or confirmed |
| | dihydropyrimidine dehydrogenase (DPD) deficiency. |
| | 7.Prior adverse reactions to anticancer therapy have not recovered to CTCAE |
| | v5.0 Grade ≤1 (excluding toxicities deemed non-risky by the investigator, |
| | such as alopecia). |
| | 8.Gastrointestinal disorders (e.g., esophageal obstruction, pyloric |
| | obstruction, intestinal obstruction), post-gastrointestinal resection, or other |
| | factors causing dysphagia that may interfere with oral drug absorption. |
| | 9.Severe comorbidities, including significant cardiac/cerebrovascular |
| | disease, uncontrolled diabetes/hypertension, active infections, or active |
| | peptic ulcer. |
| | 10.Active hepatitis B virus (HBV) infection. |
| | 11.History of immunodeficiency (e.g., HIV-positive status, |
| | congenital/acquired immunodeficiency disorders) or organ transplantation. |
| | 12.Psychiatric disorders or poor compliance. |
| | 13.Pregnancy (positive pregnancy test) or lactation. |
| | 14.Concurrent participation in another interventional clinical study or |
| | receiving other investigational therapies. |
| | 15.Concomitant use of potent CYP3A4 inhibitors/inducers or QT-prolonging |
| | drugs within 14 days prior to the first dose or during the study. |
| | 16.Other conditions deemed unsuitable for study participation by the |
| | investigator. |
| Treatment | Experimental Group |
| Regimen | Utidelone Capsules (UTD2): |

| Dosage: 50 mg/m²/day, administered orally once daily on Days 1–5. Cycle: 21 days per treatment cycle, for a total duration of 2 years. | |
|---|---|
| Cycle: 21 days per treatment cycle, for a total duration of 2 years | |
| Capecitabine: | |
| Dosage: 1000 mg/m², administered orally twice daily on Days 1–14. | |
| Cycle: 21 days per treatment cycle, for a total of 8 cycles. | |
| Treatment Discontinuation Criteria: | |
| Study treatment will be terminated if disease recurrence or intole | erable |
| adverse events (AEs) occur during the treatment period. | |
| Control Group | |
| Capecitabine: | |
| Dosage: 1000 mg/m², administered orally twice daily on Days 1–14. | |
| Cycle: 21 days per treatment cycle, for a total of 8 cycles. | |
| Treatment Discontinuation Criteria: | |
| Study treatment will be terminated if disease recurrence or intole | erable |
| adverse events (AEs) occur during the treatment period. | |
| Planned A total of 646 subjects will be enrolled, with 323 in the experimental gr | oup |
| Enrollment and 323 in the control group. | |
| Analysis Populations | |
| Full Analysis Set (FAS): Defined as all randomized subjects who me | et the |
| eligibility criteria based on the Intent-to-Treat (ITT) principle. | |
| Per Protocol Set (PPS): A subset of the FAS, excluding subjects with | major |
| protocol deviations that significantly impact the results. | |
| Safety Set (SS): Includes all randomized subjects who received at lea | st one |
| dose of the study drug. Subjects in the SS are analyzed according | to the |
| Statistical actual treatment received. | |
| Analysis Sample Size Estimation | |
| This study is a parallel-controlled superiority trial with the primary end | oint |
| being the investigator-assessed 3-year invasive disease-free survival (II | , |
| rate. Subjects are randomized 1:1 to the experimental and control group | |
| Assuming a 3-year IDFS rate of 72% in the control group and a hazard | |
| (HR) of 0.6, a total of 122 IDFS events are required to achieve 80% pov | ver at |
| a two-sided significance level of $\alpha = 0.05$ . The calculated sample size is | 418 |

subjects. Accounting for an approximate 5% dropout rate, a minimum of 440 subjects (220 per group) will be enrolled.

#### General Statistical Principles

Statistical analyses will be performed using SAS 9.4 or later. All statistical tests will be two-sided, with 95% confidence intervals (CI). Continuous data will be summarized using counts, means, standard deviations, quartiles, minima, and maxima. Categorical data will be summarized using frequencies (percentages).

### **Efficacy Analysis**

The primary endpoint, 3-year IDFS rate, will be analyzed using Kaplan-Meier survival curves with 95% CIs. The log-rank test will compare survival distributions between groups. Stratified Cox proportional hazards models will estimate HRs and 95% CIs, adjusting for postoperative pathological lymph node status. Both the FAS and PPS will be analyzed for the primary endpoint, with the FAS serving as the primary analysis set.

Overall survival (OS) will be analyzed using the same methods as IDFS. IDFS and OS rates at different timepoints will be estimated using the Kaplan-Meier method. Continuous variables will be summarized descriptively, including mean, standard deviation, median, minimum, and maximum.

#### Safety Analysis

Adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) and graded per NCI CTCAE v5.0. Safety analyses will focus on treatment-emergent AEs, treatment-related AEs, and serious AEs (SAEs). Summary tables will report the number and percentage of subjects experiencing each AE category.

# Study Duration

Patient enrollment is expected to take approximately 24 months, with the total duration of the Phase III study estimated to be 60 months.